CLINICAL TRIAL: NCT04330300
Title: The CORONAvirus Disease 2019 Angiotensin Converting Enzyme Inhibitor/Angiotensin Receptor Blocker InvestigatiON (CORONACION) Randomized Clinical Trial
Brief Title: Coronavirus (COVID-19) ACEi/ARB Investigation
Acronym: CORONACION
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Challenges with funding and very low incidence of COVID-19 at Irish study site
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Prof. John William McEvoy, Professor of Preventive Cardiology, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C.A. 2348
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Hypertension; COVID-19
Keywords: Hypertension; Blood Pressure; COVID-19; Coronavirus Disease 2019; Novel Coronavirus; Coronavirus; Cardiovascular Diseases; Pandemic; Critical Care; Intubation; Noninvasive Ventilation; Angiotensin Converting Enzyme; Angiotensin Converting Enzyme 2; Renin-Angiotensin System; Antihypertensive Agents; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Calcium Channel Blockers; Diuretics; ACE-2
MeSH Terms: conditions — Hypertension; COVID-19; Coronavirus Infections; Cardiovascular Diseases | interventions — Thiazides; Hydrochlorothiazide; Metolazone; Chlorthalidone; Chlorothiazide; Bendroflumethiazide; Indapamide; Calcium Channel Blockers; Amlodipine; Diltiazem; Felodipine; Nicardipine; Nifedipine; Nimodipine; Nitrendipine; Verapamil; Angiotensin-Converting Enzyme Inhibitors; benazepril; Captopril; Enalapril; Fosinopril; Lisinopril; Perindopril; Quinapril; Ramipril; trandolapril; Angiotensin Receptor Antagonists; candesartan; eprosartan; Irbesartan; Losartan; olmesartan; Telmisartan; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alternative anti-hypertensive medication (Experimental): Switch to an alternative BP medication (specifically a Calcium channel blocker [CCB] or Thiazide/Thiazide-like diuretic at an equipotent blood pressure lowering dose). The choice of either CCB or Thiazide/Thiazide-like anti-hypertensive provided as alternative therapy will be at the discretion of the patient's treating physician.
  Interventions: Drug: Thiazide or Thiazide-like diuretics; Drug: Calcium Channel Blockers
- Continue ACEi/ARB antihypertensive (Active Comparator): Continue with either the ACEi (Angiotensin Converting Enzyme Inhibitor) or the Angiotensin Receptor Blocker (ARB) that had already been prescribed for the treatment of hypertension.
  Interventions: Drug: ACE inhibitor; Drug: Angiotensin receptor blocker

INTERVENTIONS:
Drug: Thiazide or Thiazide-like diuretics — Anti-hypertensive (Active Arm)
  Other Names: Hydrochlorothiazide, metolazone, chlorthalidone, chlorothiazide, bendroflumethiazide, indapamide
  Arms: Alternative anti-hypertensive medication
Drug: Calcium Channel Blockers — Anti-hypertensive (Active Arm)
  Other Names: Amlodipine, diltiazem, felodipine, nicardipine, nifedipine, nimodipine, nitrendipine, verapamil
  Arms: Alternative anti-hypertensive medication
Drug: ACE inhibitor — Anti-hypertensive (Control Arm)
  Other Names: Benazepril, captopril, enalapril, fosinopril, lisinopril, perindopril, quinapril, ramipril, trandolapril
  Arms: Continue ACEi/ARB antihypertensive
Drug: Angiotensin receptor blocker — Anti-hypertensive (Control Arm)
  Other Names: Candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan
  Arms: Continue ACEi/ARB antihypertensive

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a pandemic infection caused by a virus called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Because SARS-CoV-2 is known to require the angiotensin-converting enzyme 2 (ACE-2) receptor for uptake into the human body, there have been questions about whether medications that upregulate ACE-2 receptors might increase the risk of infection and subsequent complications. One such group of medications are anti-hypertensives that block the renin-angiotensin system, including both angiotensin converting enzyme inhibitors (ACEi) and angiotensin II receptor blockers (ARB). Both ACEi and ARB are widely used for the treatment of hypertension. Early reports from China and Italy suggest that many of those who die from COVID-19 have a coexisting history of hypertension. Consequently, there have been questions raised as to whether these 2 types of blood pressure medication might increase the risk of death among patients with COVID-19. However, it is well known that the prevalence of hypertension increases linearly with age. Therefore, it is possible that the high prevalence of hypertension and ACEi/ARB use among persons who die from COVID-19 is simply confounded by age (older people are at risk of both a history of hypertension and dying from COVID-19). Whether these commonly prescribed blood pressure medications increase the risk of COVID-19 or not remains unanswered. Statements from professional cardiology societies on both sides of the Atlantic have called for urgent research into this question. Our study aims to randomize patients with primary (essential) hypertension who are already taking ACEi/ARB to either switch to an alternative BP medication or continue with the ACEi/ARB that they have already been prescribed. Adults with compelling indications for ACEi/ARB will not be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women aged 60 or over
* Known diagnosis of hypertension
* Current use of ACEi or ARB for the treatment of hypertension
* COVID-19 naïve (i.e. not known to be infected)
* English speaker

Exclusion Criteria:

* Known diabetic nephropathy
* Known heart failure with reduced ejection fraction
* Resistant hypertension (defined as blood pressure that remains above goal despite concurrent use of three anti-hypertensive agents of different classes, one of which should be a diuretic, or as blood pressure that is controlled with four or more medications)
* Contraindications or allergies to CCB or Thiazide
* Unconscious patients
* Current psychiatric in-patients
* Patients in an emergency medical setting
* Inability to consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2414 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Covid-19 positive participants who die, require intubation in ICU, or require hospitalization for non-invasive ventilation (NIV) | 12 months
  Time from randomization to the first occurrence of any of the clinical events above

SECONDARY OUTCOMES:
Number of Covid-19 positive participants who die | 12 months
  Time from randomization to the first occurrence of above
Number of Covid-19 positive participants who require intubation in intensive care unit (ICU) | 12 months
  Time from randomization to the first occurrence of above
Number of Covid-19 positive participants who require hospitalization for non-invasive ventilation (NIV) | 12 months
  Time from randomization to the first occurrence of above
Number of SARS-CoV-2 positive participants | 12 months
  Time from randomization to the first occurrence of above
Maximum troponin T value (ng/L) among Covid-19 positive participants who require acute hospitalization | 12 months
24 hour mean systolic BP (mmHg) on ambulatory BP monitoring | 12 months
  Performed in a random sub-sample of the cohort (both study arms)
All-cause mortality | 12 months
  Time from randomization to the first occurrence of above

CONTACTS AND LOCATIONS:
Overall Officials: John William McEvoy, MBBCh MHS, Principal Investigator — National University of Ireland, Galway, Ireland
Locations (1):
- University Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12-24 months
Access Criteria: To be determined